CLINICAL TRIAL: NCT02678299
Title: Phase 1/2 Study of the Combination of Pixantrone, Etoposide, Bendamustine and, in CD20 Positive Tumors, Rituximab in Patients With Relapsed Aggressive Non-Hodgkin Lymphomas of B- or T-cell Phenotype - the P[R]EBEN Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PREBEN; 2015-000758-39 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Malignant Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: PREBEN

INTERVENTIONS:
Drug: PREBEN

SUMMARY:
This is a phase 1/2 open label study to assess the safety and efficacy of pixantrone in combination with bendamustine, etoposide and , for CD20 positive B-cell lymphomas, rituximab (P[R]EBEN), in patients with relapsed aNHL of B- or T-cell phenotype.

DETAILED DESCRIPTION:
This is a phase 1/2 open label study to assess the safety and efficacy of pixantrone in combination with bendamustine, etoposide and , for CD20 positive B-cell lymphomas, rituximab (P[R]EBEN), in patients with relapsed aNHL of B- or T-cell phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed relapse of an aggressive lymphoma of T- or B-cell phenotype (including follicular lymphoma grade 3b). For excluded histological entities see 'Exclusion criteria'
* Phase 1 + Phase 2 'fit' patients:

  * Age 18-70 years at the time of inclusion
  * ECOG PS 0-1 at protocol entry
  * Deemed 'fit' by the treating physician
* Phase 2 'frail' patients:

  * Age 71-85 years at the time of inclusion and/or
  * ECOG PS 2-3 at protocol entry and/or
  * Deemed 'frail' by the treating physician
* At least six months response duration since last given course of treatment
* Estimated life expectancy of 3 months or longer
* Measurable disease
* Hemoglobin ≥ 8 g/dL (≥5 mmol/l)
* Platelets ≥ 100 x 109/L; ≥ 75 x 109/L permitted if bone marrow involvement
* Absolute neutrophil count ≥ 1.5 x 109/L; ≥ 1.0 x 109/L permitted if documented bone marrow involvement
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN); patients with proven Gilbert's syndrome (≤ 5 x ULN) may be enrolled.
* Serum glutamic-oxaloacetic transaminase (AST) and/or serum glutamic-pyruvic transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN if elevation is due to hepatic involvement by lymphoma
* Serum creatinine ≤ 2 x ULNb
* Women of childbearing potential must use safe anticonception (e.g. contraceptive pills, intrauterine devices etc.) during the study and 12 months after the last administration of study drugs
* Male patients must use contraception for the duration of the study and 6 months after the last administration of study drugs if his partner is of childbearing potential
* Written informed consent

Exclusion Criteria:

* Patients with primary refractory disease (e.g. progressing under platinum-containing or similar salvage therapy) defined as < 6 months response duration from last given course of treatment.
* High-dose therapy with autologous stem cell rescue within the last 6 months prior to study entry.
* Following T-cell lymphoma entities:

  * T-cell lymphoblastic lymphoma
  * Hepatosplenic T-cell lymphoma
  * Extranodal NK/T, nasal type
  * Subcutaneous panniculitis-like
  * Primary cutaneous T-cell lymphoma
  * Primary leukemic T-cell lymphoma
* Following B-cell lymphoma entities:

  * Transformed indolent B-cell lymphomas
  * Post-transplant B-cell lymphoproliferative disease
  * HIV-associated B-cell lymphoma
* Concurrent severe and/or uncontrolled medical disease which is not lymphoma-related
* Left ventricular ejection fraction (LVEF) < 45%
* Suspected or documented central nervous system involvement by NHL
* Patients known to be antigen positive for HIV and/or hepatitis B and/or hepatitis C
* Patients with active, uncontrolled infections
* Vaccination with live, attenuated vaccines within 4 weeks of inclusion
* Pregnant and/or breastfeeding women
* History of active cancer during the past 5 years, except basal carcinoma of the skin or stage 0 cervical carcinoma
* Known hypersensitivity to one or more of the study drugs
* Unwillingness or inability to comply with the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2022-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MTD of pixantrone, bendamustine and etoposide in 'fit' relapsed aNHL pts (phase 1) | 1.5 yrs
Objective ORR in both 'fit' and 'frail' relapsed aNHL pts (phase 2) | 4 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Francesco d'Amore, MD DMSci, Principal Investigator — Dept. of Hematology, Aarhus University Hospital
Locations (18):
- Denmark (3):
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Department of Hematology, Copenhagen University Hospital, Copenhagen
  - Department of Hematology, Odense University Hospital, Odense
- Helsinki University Hospital Comprehensive Cancer Center, Helsinki, Finland
- Netherlands (10):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Meander Medical Center, Amersfoort
  - Slingeland Hospital, Doetinchem
  - Albert Schweitzer Hospital, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Hospital, Flushing
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Ziekenhuis, Hoofddorp
  - Erasmus Medical Center, Rotterdam
  - Haga Hospital, loc. Leyweg, The Hague
- Norway (3):
  - Department of Oncology, Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Department of Oncology, St. Olavs Hospital, Trondheim
- Department of Oncology, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No